CLINICAL TRIAL: NCT02321254
Title: A Pilot Study of Active, Robot-assisted Therapy for Shoulder Rehabilitation After Stroke, Using Myoelectric Signals
Brief Title: Myoelectric Robot-assisted Rehabilitation for the Upper Limb After Stroke
Acronym: MyoReArm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Collaborators: FerRobotics Compliant Robot GmbH, Linz, Austria (Unknown)
Responsible Party: Principal Investigator, Andrea Turolla, Head of Laboratory of Kinematics and Robotics, IRCCS San Camillo, Venezia, Italy
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Prot.2013.16
Record Dates: First submitted 2014-12-11; First posted 2014-12-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Stroke
Keywords: Stroke; Upper limb; Robotics; Electromyography; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- The RehaARM-Robot (Experimental): Receive 45 min of robot-assisted therapy for the shoulder and 1 hour of daily standard rehabilitation therapy.
  Interventions: Device: The RehaARM-Robot; Behavioral: Standard rehabilitation therapy

INTERVENTIONS:
Device: The RehaARM-Robot — Robot therapy by using a 3-Degrees-Of-Freedom (3DOFs) robot to train the shoulder.
  Other Names: Robot-assisted therapy for the shoulder
Behavioral: Standard rehabilitation therapy — Standard therapy of stroke rehabilitation including speech, physical, occupational therapies and group activities.

SUMMARY:
The aim of this study is to assess the clinical effectiveness of the RehaARM-robot and to determine the feasibility of including robotic therapy in daily rehabilitation programmes, after stroke. Additionally, we aim to investigate the acceptance of this intervention from patients and therapists. A total of 10 patients will be recruited in this study, all the patients will receive 1 hour of standard therapy together with 45 min of robot therapy every day. The robot therapy will last 45 minutes, for 15 consecutive days within a maximum period of four weeks. Additional 15 minutes are required for placing surface electrodes on the shoulder and patient preparation. The study will include passive and active shoulder training of four movements: Horizontal abduction/adduction, abduction/adduction, internal/external rotation and flexion/extension. The passive part lasts 10 minutes and the active part 35 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from stroke, ischemic and / or hemorrhagic
* Stroke in the left hemisphere
* Score between 1 and 3 in the upper-limb sub-item of the Italian version of the National Institute of Health Stroke Scale (IT-NIHSS) (Pezzella et al. 2009)
* Score of the Functional Independence Measure (FIM) scale (Keith et al., 1987) less than 100 out of a total of 126. This scale is used as a reference to indicate the degree of autonomy in carrying out activities of daily living (ADLs)
* Score of the upper-limb Fugl-Meyer scale (FMA) (Fugl-Meyer et al., 1975) less than 60. This scale measures the residual motor function of a person after stroke

Exclusion Criteria:

* Non-stabilized fractures
* Diagnosis of depression
* Traumatic brain Injury
* Pharmacologically uncontrolled epilepsy
* Ideomotor apraxia
* Neglect
* Mini Mental State Examination (MMSE) score <20/30
* Severe impairment of verbal comprehension, defined by a score in the Token Test (Tau points<58/78)
* Patients participating in other rehabilitation treatments for the upper-limb (e.g. virtual reality treatment, motor imagery, etc)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment scale - Upper Extremity (FMA-UE) | 3 weeks (15 sessions)
  Motor function of the upper limb is measured by means of the Upper Extremity Motor Assessment of the Fugl-Meyer Assessment Scale.

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) | 3 weeks (15 sessions)
  FIM is an 18-item scale that assesses patient's disability and medical rehabilitation functional outcome (A total of 126 points).
Reaching Performance Scale (RPS) | 3 weeks (15 sessions)
  It assesses the ability of subjects to reach an object (a cone). The cone is placed at a 4-cm distance and after at a 30-cm distance from the subject. The subject is asked to reach and grab the cone if possible. The observer evaluates the quality of reaching instead of the grip strength ( A total of 36 points).
Modified Ashworth Scale (MAS) of five muscles | 3 weeks (15 sessions)
  Spasticity is measured using the MAS of five muscles: Pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus (Total of 20 points).
Nine Hole Pegboard Test (NHPT) | 3 weeks (15 sessions)
  It measures the dexterity of the hand. Patient should insert 9 pins in the board. There are 9 pins. The number of pins inserted in 50 min are registered or if the patient inserted 9 pins, then the time is registered.

OTHER OUTCOMES:
Shoulder active range of movement (ROM-S) | 3 weeks (15 sessions)
  Active range improvement for shoulder abduction and flexion are measured using the Tyromotion Pablo System.
• Average amount of active task repetitions of a sequence of motor tasks using the robot during a 1-hour therapy treatment. | 3 weeks (15 sessions)
  A higher number of repetitions is a paramount for neuroplasticity. The ability of subjects to execute a larger of number of motor task repetitions with the robot after the treatment is measured.
• Smoothness of the torque (i.e. Number of peaks of the torque, [n]) for a sequence of motor tasks using the robot during a 1-hour therapy treatment . | 3 weeks (15 sessions)
  Smoothness is a measure of human movement coordination. Improvement of smoothness after the treatment is measured.
• Average magnitude of the muscle activation during the active phase normalized by duration of the active phase (magnitude/time) for a sequence of motor tasks using the robot during a 1-hour therapy treatment. | 3 weeks (15 sessions)
• Average similarity between the muscle (synergy) modules of the paretic arm and the muscle modules of the right arm of healthy subjects for a standard sequence of motor tasks using the robot during a 1-hour therapy treatment | 3 weeks (15 sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Turolla, MSc, Principal Investigator — IRCCS San Camillo Hospital Foundation, Venice (Italy)
Locations (2):
- FerRobotics Compliant Robot Technology GmbH, Linz, Austria
- IRCCS San Camillo Hospital Foundation, Venice, Italy

REFERENCES:
- [Result] Liao WW, Wu CY, Hsieh YW, Lin KC, Chang WY. Effects of robot-assisted upper limb rehabilitation on daily function and real-world arm activity in patients with chronic stroke: a randomized controlled trial. Clin Rehabil. 2012 Feb;26(2):111-20. doi: 10.1177/0269215511416383. Epub 2011 Aug 12. PMID 21840917
- [Result] Suputtitada A, Suwanwela NC, Tumvitee S. Effectiveness of constraint-induced movement therapy in chronic stroke patients. J Med Assoc Thai. 2004 Dec;87(12):1482-90. PMID 15822545
- [Result] Makowski NS, Knutson JS, Chae J, Crago PE. Functional electrical stimulation to augment poststroke reach and hand opening in the presence of voluntary effort: a pilot study. Neurorehabil Neural Repair. 2014 Mar-Apr;28(3):241-9. doi: 10.1177/1545968313505913. Epub 2013 Nov 22. PMID 24270058
- [Result] Mehrholz J, Hadrich A, Platz T, Kugler J, Pohl M. Electromechanical and robot-assisted arm training for improving generic activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2012 Jun 13;(6):CD006876. doi: 10.1002/14651858.CD006876.pub3. PMID 22696362
- [Result] Laver KE, George S, Thomas S, Deutsch JE, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008349. doi: 10.1002/14651858.CD008349.pub2. PMID 21901720
- [Result] Turolla A, Dam M, Ventura L, Tonin P, Agostini M, Zucconi C, Kiper P, Cagnin A, Piron L. Virtual reality for the rehabilitation of the upper limb motor function after stroke: a prospective controlled trial. J Neuroeng Rehabil. 2013 Aug 1;10:85. doi: 10.1186/1743-0003-10-85. PMID 23914733
- [Result] Kwakkel G, Kollen BJ, Krebs HI. Effects of robot-assisted therapy on upper limb recovery after stroke: a systematic review. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):111-21. doi: 10.1177/1545968307305457. Epub 2007 Sep 17. PMID 17876068
- [Result] Johansson BB. Current trends in stroke rehabilitation. A review with focus on brain plasticity. Acta Neurol Scand. 2011 Mar;123(3):147-59. doi: 10.1111/j.1600-0404.2010.01417.x. Epub 2010 Aug 19. PMID 20726844
- [Result] Hermens HJ, Freriks B, Disselhorst-Klug C, Rau G. Development of recommendations for SEMG sensors and sensor placement procedures. J Electromyogr Kinesiol. 2000 Oct;10(5):361-74. doi: 10.1016/s1050-6411(00)00027-4. PMID 11018445
- [Result] Sartori M, Reggiani M, Farina D, Lloyd DG. EMG-driven forward-dynamic estimation of muscle force and joint moment about multiple degrees of freedom in the human lower extremity. PLoS One. 2012;7(12):e52618. doi: 10.1371/journal.pone.0052618. Epub 2012 Dec 26. PMID 23300725